CLINICAL TRIAL: NCT04756466
Title: Multicenter, Randomized, Double-blind Parallel Group Pilot Study to Evaluate the Effect of the Consumption of a Lactobacillus Strain on the Incidence of Covid-19 in the Elderly
Brief Title: Effect of the Consumption of a Lactobacillus Strain on the Incidence of Covid-19 in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P055
Record Dates: First submitted 2021-01-21; First posted 2021-02-16 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: SARS CoV-2 Infection; Elderly
Keywords: Probiotics; COVID19
MeSH Terms: conditions — COVID-19 | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group that will receive a daily placebo capsule consisting of maltodextrin during 3 months
  Interventions: Dietary Supplement: Placebo
- Probiotic group (Experimental): Experimental group that will receive one capsule with the probiotic strain per day (3x10 9 CFU / day) during 3 months
  Interventions: Dietary Supplement: Lactobacillus

INTERVENTIONS:
Dietary Supplement: Placebo — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Control group
Dietary Supplement: Lactobacillus — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Probiotic group

SUMMARY:
The objective of this trial is to evaluate the effect of the consumption of a probiotic strain on the incidence and severity of COVID-19 in elderly population living in a nursing home. In addition, it will be evaluated if the probiotic strain have some effect on the immune response generated by the Covid-19 vaccine inthis population.

DETAILED DESCRIPTION:
The working hypothesis is that the administration of a Lactobacillus strain improves the immune response in the elderly population, improving the immune response to a possible COVID-19 infection. The strain would act as an adjuvant that contributes to developing an effective response against the virus, and therefore there are fewer infectious symptoms due to this virus or, if it appears, it occurs in a milder way among the subjects who take the probiotic strain. Also,the investigators hypothesizes that the administration of the Lactobacillus may improve the immune response generated by the Covid-19 vaccine in this elderly population.

ELIGIBILITY:
Inclusion Criteria:

1. Person over 60 years of age.
2. Intern in residence for the elderly.
3. Sign informed consent.

Exclusion Criteria:

1. Person who at some previous time has tested positive for detection of COVID-19 by PCR or serology.
2. Person who at the time of starting the intervention presents symptoms compatible with COVID-19.
3. Person with concomitant disease type HIV, transplant, active cancer or other type of active immunosuppression.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS CoV-2 infection. | 3 months
  Incidence of SARS CoV-2 infection confirmed by PCR or antigen test

SECONDARY OUTCOMES:
Incidence of hospital admissions caused by SARS-CoV-2 infection . | 3 months
  Incidence of hospital admissions caused by infection caused by SARS-CoV-2 confirmed by PCR or antigen test
Incidence of ICU admissions caused by SARS-CoV-2 infection | 3 months
  Incidence of ICU admissions caused by infection caused by SARS-CoV-2 confirmed by PCR or antigen test
Incidence of pneumonia caused by SARS-CoV-2 infection . | 3 months
  Incidence of pneumonia caused by infection caused by SARS-CoV-2 confirmed by PCR or antigen test
Incidence of need for oxygen support due to SARS-CoV-2 infection.. | 3 months
  Incidence of need for oxygen support due to SARS-CoV-2 infection confirmed by PCR or antigen test.
Incidence of gastrointestinal symptoms due to SARS-CoV-2 infection. | 3 months
  Incidence of gastrointestinal symptoms due to SARS-CoV-2 infection confirmed by PCR or antigen test.
Days with body temperature> 37.5ºC. | 3 months
  In case of SARS-CoV-2 infection confirmed by PCR or antigen test, Days with body temperature> 37.5ºC
Days of persistent cough. | 3 months
  In case of SARS-CoV-2 infection confirmed by PCR or antigen test, Days with persistent cough
Days of persistent feeling of fatigue. | 3 months
  In case of SARS-CoV-2 infection confirmed by PCR or antigen test, Days of persistent feeling of fatigue.
Use of pharmacological treatments. | 3 months
  In case of SARS-CoV-2 infection confirmed by PCR or antigen test, use of pharmacological treatments
Serum levels of IgG antibody against SARS-CoV-2 | 6-weeks from second dose of the vaccine
  In case volunteers was vaccinated against SARS-CoV-2, the serum levels of IgG antibody against SARS-CoV-2 will be measured, at 6 weeks from the second dose of the vaccine
Serum levels of IgA antibody against SARS-CoV-2 | 6-weeks from second dose of the vaccine
  In case volunteers was vaccinated against SARS-CoV-2, the serum levels of IgA antibody against SARS-CoV-2 will be measured, at 6 weeks from the second dose of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Olivares, PhD, Study Director — Biosearch S.A.; Anxo Fernandez-Ferreiro, PhD, Principal Investigator — Complejo Hospitalario Universitario de Santiago Compostela
Locations (3):
- Spain (3):
  - Residencia San Marcos, Santiago de Compostela, A Coruña
  - Residencia Santa Olalla, Santiago de Compostela, A Coruña
  - Residencia San Simon de Ons, Santiago de Compostela, A Coruña

IPD SHARING:
Plan to Share IPD: No